CLINICAL TRIAL: NCT03789097
Title: In Situ Vaccination With Flt3L, Radiation, and Poly-ICLC Combined With Pembrolizumab in Patients With Non-Hodgkin's Lymphoma, Metastatic Breast Cancer, and Head and Neck Squamous Cell Carcinoma
Brief Title: Vaccination With Flt3L, Radiation, and Poly-ICLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celldex Therapeutics (Industry)
Responsible Party: Principal Investigator, Joshua Brody, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 19-0477; GCO 18-2394 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Non-Hodgkin's Lymphoma; Metastatic Breast Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: Radiation; Poly-ICLC; Pembrolizumab; Lymphoma; Breast Cancer; Carcinoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Lymphoma; Carcinoma | interventions — pembrolizumab; Radiation; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination therapy (Experimental): Vaccination with Flt3L, Radiation, and Poly ICLC combined with Pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Flt3L; Radiation: Radiation; Drug: Poly ICLC

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg administered as an IV infusion over 30 minutes Q3W
  Other Names: Keytruda
Drug: Flt3L — an immune cell growth factor. CDX-301 drug product is formulated as a sterile solution intended for single-use parenteral administration. Each vial contains a nominal 2.5 mg/mL CDX-301 protein in a 1 mL volume of buffered solution composed of sodium phosphate and sodium chloride, with a pH of 7.0.
  Other Names: CDX-301; Recombinant Human Flt3 Ligand
Radiation: Radiation — The target site will get 2 small treatments of radiation.
Drug: Poly ICLC — an immune cell activating factor. vials containing 1 ml of 2 mg/mL
  Other Names: Hiltonol

SUMMARY:
This is a combination of 4 therapies, three of which are used to treat a single "target site" of your cancer (such as a lymph node or a single tumor), and the 4th is given directly into the blood stream (intravenous or "IV").

1. Radiation: The target site --lymph node or tumor (the one what will be injected) --will get two small treatments of radiation. Radiation is often times used to shrink and kill tumors in patients with certain types of lymphoma, breast cancer and head and neck cancer, however, the dose of radiation that you will receive --one dose on day one of the clinical trial and one dose on day two --is 10 to 20 time less radiation that you would receive for treatment of these cancers.
2. Flt3L/CDX-301 is an immune cell growth factor, similar to white blood cell growth factors (Neupogen or Neulasta) or red blood cell growth factors (EPO or Epogen) that you may have received to help protect your blood cells previously. Flt3L causes your body to make more immune cells, specifically a type of immune cell called "dendritic cells".
3. Poly-ICLC is an immune cell activating factor. Its function is to turn on the immune cells that have been brought to the tumor by Flt3L.
4. Pembrolizumab is an antibody (a type of human protein) that is being tested to see if it will allow the body's immune system to kill your tumor cells. Pembrolizumab is approved for use by the U.S. Food and Drug Administration (FDA) for the treatment of adult patients with many different types of cancer including head and neck cancer. Pembrolizumab is not FDA approved to treat patients with non-Hodgkin's lymphoma or metastatic breast cancer, as it has not been effective at treating these cancers when used alone. While most people do not have immediate side effects when this medication is given, it has the ability to cause side effects for.

DETAILED DESCRIPTION:
Phase 1 and Phase 2 will occur sequentially:

Phase 1 is the preliminary safety assessment portion of the study, which will follow a modified 3 + 3 design to assess toxicity. The trial would be held for review should there be more than 1 dose-limiting toxicity (DLT) observed within the first 3-6 patients. The toxicity of the in situ vaccine without pembrolizumab (ongoing and previous trials) has been minimal, limited to transient febrile response to the intratumoral Toll-like receptor (TLR) ligand poly-ICLC, typically resolving with oral acetaminophen. As such, the primary objective of Phase 1 is to assess the safety of the addition of pembrolizumab to this in situ vaccine protocol. In Phase 1, patients will only be enrolled at the lead institution (Mount Sinai). After enrollment of the initial 3 patients, enrollment will pause until all three patients have completed cycle 1 of pembrolizumab (DLT evaluation window is 63 days from initiation of in situ vaccine). During the pause, new patients may be consented and screened, but not initiated on therapy. If 1 or no DLTs are observed in the first 3 patients, an additional 3 patients will be enrolled. The regimen will be considered safe (in order to progress to Phase 2) if no more than 1 out of 6 patients experience a DLT. If two or more DLTs are observed at any point in Phase 1 then accrual will be stopped for protocol review by Data Safety Monitoring Board, PIs and sponsor for possibility of protocol amendment.

Phase 2 will follow a Simon's two-stage design. This Phase will proceed only if toxicity is acceptable as determined in Phase 1.

Phase 1/2 design: Patients will be enrolled concurrently into three independent cohorts, with patients from Phase 1 evaluated within their subsequent disease-specific cohorts. iNHL, MBC and HNSCC often have peripherally accessible tumors amenable to intratumoral injection, and have all had relatively modest responses to single-agent checkpoint blockade, so are good candidates for this novel combination. Patients will be enrolled regardless of the PD-L1 staining of their tumor. We will also enroll patients previously exposed to PD-1/PD-L1 targeted therapies either on a clinical trial or as standard of care (as for HNSCC).

Cohort A: iNHL including but not limited to chronic lymphocytic leukemia (CLL/SLL), follicular lymphoma (FL), and marginal zone lymphoma (MZL). This cohort excludes patients with diffuse large B cell lymphoma (DLBCL) and any other lymphoma determined to be progressing rapidly by investigator (PI or site PI).

Cohort B: MBC with peripherally palpable disease amenable to intratumoral injection.

Cohort C: HNSCC with peripherally palpable disease amenable to intratumoral injection.

Stage 1: Seven patients will be evaluated in Stage 1 of Phase 2 in each disease-specific cohort, inclusive of patients enrolled in Phase 1. If no patient in a cohort achieves a response, the study in that cohort will close due to a lack of efficacy. The first seven patients in each histology will only be enrolled at Mount Sinai.

Stage 2: If one or more responses are seen in Stage 1, enrollment of an additional 12 patients for Cohorts A and B or 11 patients for Cohort C will proceed. These cohorts may be also be enrolled at collaborator sites (to be determined).

* Cohorts A or B: If at least three out of the 19 patients achieve a response, the intervention will be considered promising and worthy of further investigation.
* Cohort C: If at least four out of the 18 patients achieve a response, the intervention will be considered promising and worthy of further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Have pathologically confirmed iNHL, MBC or HNSCC
* Lymphoma subtypes that may be enrolled include small lymphocytic lymphoma

Exclusion Criteria:

* Is currently participating and receiving an investigational therapy (not standard therapies) or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days of the first dose of treatment.
* Any patients that require immediate treatment or cytoreduction are excluded. Note: This is applicable for iNHL, MBC, and HNSCC populations.
* Any patient with transformed lymphoma, or patients with grade 3A follicular lymphoma are excluded.
* MZL patients with gastric MALT lymphomas with disease localized to the stomach are excluded, and any patient with disease in a site where injection is determined to be high risk.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
* Hypersensitivity to pembrolizumab, poly-ICLC, Flt3L or any of their excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 28 days prior to study D22 (First dose of pembrolizumab) or who has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to agents administered more than 28 days before initiation of in situ vaccine protocol.
* Has had prior chemotherapy, targeted small molecule therapy, or RT therapy within 14 days prior to study D0 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to a previously administered agent. Note: Patients with chronic ≤ Grade 2 AEs such as neuropathy are an exception to this criterion and may qualify for the study.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has known active central nervous system metastases, leptomeningeal disease and/or lymphomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 28 days prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include leptomeningeal disease or lymphomatous meningitis, which are excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a systemic treatment. Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy at time of enrollment in trial.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical or anal cancer, prostate cancer on stable dose of hormonal therapy without rising PSA.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Has known psychiatric or substance abuse disorders that investigator believes would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment (roughly two and a half years after enrollment).
* HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen.
* Has known active Hepatitis B (e.g., HBV detected by PCR) or active Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Patients with grade 3B follicular lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 63 days
  DLTs recorded and graded according to NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.03, within DLT evaluation window of 63 days (end of cycle 1 of pembrolizumab) from initiation of in situ vaccine.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 months
  Overall response rate (ORR) as defined as best response achieved within the first 6 months from initiation of trial. ORR is defined as complete remission (CR) or partial remission (PR) in patients as defined by RECIST v1.1 for MBC and HNSCC or as per the RECIL Criteria for patients with lymphoma, determined by Positron emission tomography-computed tomography (PET/CT) or computed tomography (CT) imaging which occurs at 3 month intervals, with the first imaging 3 months following initiation of Flt3L (D0) +/- 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Brody, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States